CLINICAL TRIAL: NCT04398810
Title: A Comparison of Postoperative Pain Results According to Pressure to Form Pneumoperitoneum During Robot-assisted Single-port Cholecystectomy; a Randomized Controlled Trial.
Brief Title: Postoperative Pain Results According to Pressure to Form Pneumoperitoneum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul-09
Record Dates: First submitted 2020-05-12; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Cholecystitis; Postoperative Pain
Keywords: robot cholecystectomy; low-pressure pneumoperitoneum; postoperative pain
MeSH Terms: conditions — Cholecystitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the low-pressure pneumoperitoneum during surgery (Experimental): A. Inclusion criteria Patients who underwent elective gallbladder surgery
  * Cholelithiasis
  * Chronic cholecystitis
  * Gallbladder polyps
  * Gallbladder adenoma
  * Porcelain gallbladder
  The experimental group controls the CO2 flow that is injected into the abdominal cavity during surgery and maintains the pressure in the abdominal cavity at a low level of 5 mmHg to perform the surgery.
  Interventions: Procedure: robotic single port cholecystectomy
- the standard-pressure pneumoperitoneum during surgery (Experimental): A. Inclusion criteria Patients who underwent elective gallbladder surgery
  * Cholelithiasis
  * Chronic cholecystitis
  * Gallbladder polyps
  * Gallbladder adenoma
  * Porcelain gallbladder
  In the case of the control group, surgery is performed while maintaining the pressure in the abdominal cavity at 12 mmHg as generally performed during surgery.
  Interventions: Procedure: robotic single port cholecystectomy

INTERVENTIONS:
Procedure: robotic single port cholecystectomy — 1. Local anesthetic administration during wound incision In the experimental group and the control group, a local anesthetic was administered to the wound surface when a glove port was installed on the navel at the start of surgery. (bupivacaine 0.5% 14ml subcutaneous injection)
  2. Residual gas aspiration
  3. Pulmonary recruitment maneuver In both the experimental group and the control group, before the operation was completed and the wound was closed, the patient was taken to the Trenedelenburg position, and then the pressure of 60 cm H2o in the abdomen was applied, and manual inflation was performed twice, 5 seconds at a time, and pulmonary recruitment was performed.
  4. Warming of the washing solution in the abdominal cavity

SUMMARY:
This study showed the difference in postoperative pain between the groups that performed surgery with the low-pressure pneumoperitoneum and the group that performed surgery in the standard-pressure pneumoperitoneum when robotic single-hole cholecystectomy was performed.

The primary purpose of the study was to compare the differences in the visual analog scale (VAS) between the two groups and to demonstrate the effectiveness of pain relief after surgery.

Secondly, the effect of the low-pressure pneumoperitoneum on the patient's postoperative recovery and outcome was compared with the control group by comparing the length of stay, operation time, and postoperative complications.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy was the most common treatment method for gallbladder-related diseases, and robotic cholecystectomy was also currently being performed. Many patients complained pain around the wound, shoulder and back after surgery. Several methods had been attempted to reduce postoperative pain, previous studies showed that oral medications such as NSAIDS, administration of local anesthetics in wounds and abdominal cavity, low-pressure penumoperitoneum, humidification of intraperitoneal washing fluid, And active residual gas suction in the abdominal cavity had been found to relieve postoperative pain.

Robotic cholecystectomy, similar to laparoscopic cholecystectomy, also formed pneumoperitoneum to secure the surgical space during operation. Based on the results published in various studies, it had known that the most effective method of pain relief for laparoscopic pain was to create low-pressure pneumoperitoneum.

In this study, investigators attempted to prove the effectiveness of low pressure pneumoperioneum through a prospective randomized controlled trial between the experimental group with the low-pressure pneumoperitoneum and the control group with the standard-pressure pneumoperitoneum during robotic single-hole cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent elective gallbladder surgery

* Cholelithiasis
* Chronic cholecystitis
* Gallbladder polyps
* Gallbladder adenoma
* Porcelain gallbladder

Exclusion Criteria:

1. Acute cholecystitis patient group

   * Necrotic gallbladder
   * Collapsed gallbladder
   * Gallbladder pustosis
   * Gallbladder emphysema
   * Hemorrhagic gallbladder
   * Perforated gallbladder
2. cholecystitis with a gallbladder thickness of 4 mm or more on CT or ultrasound
3. cholecystitis with adhesions to surrounding organs due to inflammation of the gallbladder
4. Patient group performing surgery concurrently due to other organ diseases
5. Immunosuppressive patient group

   * Transplant patient group: Liver transplant patient group (PSLT), Kidney transplant patient group (PSKT)
   * AIDS patients group
6. Patient group with history of open abdominal surgery
7. Transplant group during open surgery
8. Patients under 19 years of age.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-06-02 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score(VAS) | 24 hours after surgery
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.

SECONDARY OUTCOMES:
postoperative complication | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  postoperative complication : bile leakage, atelectasis, pneumonia, wound infection, bleeding, etc..
hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  hospital stay(days) : The duration between the operation day and the day of discharge
operation time | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  operation time(minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Won jong Kim, MD, Study Director — The Catholic University of Korea
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: No